CLINICAL TRIAL: NCT00948493
Title: An Open-Label Treatment Investigational New Drug (IND) for the Use of Generex Oral-lyn™ in Patients With Type 1 or Type 2 Diabetes Mellitus
Brief Title: Treatment Use of Generex Oral-lyn™ in Patients With Diabetes
Status: No longer available | Type: Expanded Access
Sponsor: Generex Biotechnology Corp. (Industry)
Responsible Party: Sponsor
Other Study IDs: GEN-100-OL
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: diabetes; insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

INTERVENTIONS:
Drug: Buccal insulin spray — Oral insulin spray absorbed in buccal mucosa
  Other Names: Generex Oral-lynTM (oral, buccal insulin spray)

SUMMARY:
The objective of this Treatment IND protocol is to provide Generex Oral-lyn™ to patients with serious or life-threatening Type 1 or Type 2 diabetes mellitus, with no satisfactory alternative therapy available for treatment of diabetes, and who are not eligible to participate in the ongoing pivotal clinical trial (Protocol GEN-084-OL). This protocol is intended as a substitute for the Single Patient IND mechanism to obtain Generex Oral-lyn™.

ELIGIBILITY:
Study is closed

Sex: All
Age Groups: Child, Adult, Older Adult